CLINICAL TRIAL: NCT05316038
Title: Study of the Impact of Belatacept Conversion on Metabolic and Infectious Complications in Kidney Transplant Recipients at Grenoble-Alpes University Hospital
Brief Title: Metabolic and Infectious Complications Post Belatacept Conversion
Acronym: Belaswitch
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, EssaiClinique_Belaswitch, Pincipal investigator, University Hospital, Grenoble
Other Study IDs: Belaswitch_Grenoble
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Kidney Transplant Infection; Cardiovascular Diseases; Immunosuppression; Kidney Transplant; Complications
Keywords: transplantation; Belatacept; TTV; Cardio-vascular complications
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood mononucleated cell Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Belatacept cohort: Kidney transplanted patients for whom a conversion from Tacrolimus to belatacept has been decided will be included in this cohort.
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — The test is performed on an empty stomach for at least 10 hours. The first blood sugar level is taken on an empty stomach. Then ingestion of 75g of sugar. A second blood test takes place 1 hour after the sugar intake and the third blood sugar test takes place 2 hours after the sugar intake.

SUMMARY:
The BELASWITCH study is a prospective single-centre study including all kidney transplant patients for whom a conversion from Tacrolimus to Belatacept has been decided by the transplant clinicians of the Grenoble Alpes University Hospital.

Each patient will be included at the time of conversion (patients stable on Tacrolimus for at least 6 months) and will be their own control 1 year after conversion to Belatacept.

The study has two components:

* A "Metabolic" benefit arm: the investigators assume that conversion from Tacrolimus to Belatacept reduces the risk of diabetes by reducing the level of insulin resistance.
* An "Infectious" risk arm: measurement of the viral load of Torque Teno Virus to assess the state of immunosuppression of patients. In this sense, the investigators hypothesise that it could serve as a biomarker of immunodepression in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have had a kidney transplant more than 6 months ago.
* Whose immunosuppression includes stable Tacrolimus (change in dose or dosage form allowed) for at least 3 months.
* Therapeutic plan to change Tacrolimus-based immunosuppression to Belatacept
* Having signed the consent of collection CRB04 - Nephrology Collection (last authorization number: AC-2019-3627) and the BELASWITCH protocol consent.

Exclusion Criteria:

* Subjects under guardianship or deprived of liberty
* Patients who object to the use of their data and/or samples in the research
* Patients having received an immunosuppressive treatment different from the standard one (Tacrolimus, mycophenolate mofetil or Everolimus, corticosteroids)
* ABO and/or HLA incompatible kidney transplantation

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The BELASWITCH study cohort is a prospective single-centre study including all adult kidney transplant recipients for whom a conversion from Tacrolimus to Belatacept has been decided by the transplant clinicians of the Grenoble Alpes University Hospital.
  Each patient will be included at the time of conversion (patients stable on Tacrolimus for at least 6 months) and will be their own control 1 year after conversion to Belatacept.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Oral glucose tolerance test results in kidney transplant patients on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 1 year | 1 year
Torque TenoVirus replication (in copies/ml) in kidney transplant patients on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year. | 1 year

SECONDARY OUTCOMES:
Comparison of weight and height (combined to report BMI in kg/m^2) on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year | 1 year
Comparison of blood pressure in mmHg on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year | 1 year
Comparison of abdominal perimeter of kidney transplant recipients in centimeters on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year | 1 year
Comparison of HbA1c measurment in percentage on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year | 1 year
Comparison of LDL measurment in g/l on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year | 1 year
Comparison of HDL measurment in g/l on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year | 1 year
Comparison of triglycerides measurment in g/l on Tacrolimus (M-1 and D0) and after conversion to Belatacept at 3 months, 6 months and 1 year | 1 year
Number of major cardiovascular events (stroke, coronary syndrome, hospitalization for cardiac decompensation, death from cardiovascular causes) | 1 year
Correlation of TorqueTenoVirus replication in copies/ml with the occurrence of opportunistic infections (Cytomegalovirus, Epstein-Barr virus, BKVirus). | 1 year
  Opportunistic infections are defined as positive DNAemia in copies/ml
Correlatation of TorqueTenoVirus replication (in copies/ml) with immunosuppressant assays: Tacrolimus (µg/l) at M-1 and D0 and Belatacept (µg/l) at M3, M6 and M12 | 1 year
Correlation of TorqueTenoVirus in copies/ml and the risk of biopsy-proven renal transplant rejection up to M12 after conversion to Belatacept. | 1 year
  Rejection are defined according to the more recent histological Banff classification
Compare the performance of TorqueTenoVirus quantitative polymerase chain reaction in copies/ml performed on plasma and whole blood samples | 3 months
Trough Plasma Concentration of Belatacept | 3 months
Area under the plasma concentration versus time curve (AUC) of Belatacept | 3 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Collins AJ, Foley RN, Gilbertson DT, Chen SC. United States Renal Data System public health surveillance of chronic kidney disease and end-stage renal disease. Kidney Int Suppl (2011). 2015 Jun;5(1):2-7. doi: 10.1038/kisup.2015.2. PMID 26097778
- [Result] Dharnidharka VR. Costimulation blockade with belatacept in renal transplantation. N Engl J Med. 2005 Nov 10;353(19):2085-6; author reply 2085-6. doi: 10.1056/NEJM200511103531919. No abstract available. PMID 16282187
- [Result] Vincenti F, Rostaing L, Grinyo J, Rice K, Steinberg S, Gaite L, Moal MC, Mondragon-Ramirez GA, Kothari J, Polinsky MS, Meier-Kriesche HU, Munier S, Larsen CP. Belatacept and Long-Term Outcomes in Kidney Transplantation. N Engl J Med. 2016 Jan 28;374(4):333-43. doi: 10.1056/NEJMoa1506027. PMID 26816011
- [Result] Durrbach A, Pestana JM, Florman S, Del Carmen Rial M, Rostaing L, Kuypers D, Matas A, Wekerle T, Polinsky M, Meier-Kriesche HU, Munier S, Grinyo JM. Long-Term Outcomes in Belatacept- Versus Cyclosporine-Treated Recipients of Extended Criteria Donor Kidneys: Final Results From BENEFIT-EXT, a Phase III Randomized Study. Am J Transplant. 2016 Nov;16(11):3192-3201. doi: 10.1111/ajt.13830. Epub 2016 Jun 9. PMID 27130868
- [Result] Baron PW, Infante S, Peters R, Tilahun J, Weissman J, Delgado L, Kore AH, Beeson WL, de Vera ME. Post-Transplant Diabetes Mellitus After Kidney Transplant in Hispanics and Caucasians Treated with Tacrolimus-Based Immunosuppression. Ann Transplant. 2017 May 23;22:309-314. doi: 10.12659/aot.903079. PMID 28533501
- [Result] Iida S, Ishida H, Tokumoto T, Omoto K, Shirakawa H, Shimizu T, Amano H, Setoguchi K, Nozaki T, Toki D, Tokita D, Tanabe K. New-onset diabetes after transplantation in tacrolimus-treated, living kidney transplantation: long-term impact and utility of the pre-transplant OGTT. Int Urol Nephrol. 2010 Dec;42(4):935-45. doi: 10.1007/s11255-010-9712-0. Epub 2010 Feb 19. PMID 20169408
- [Result] Drachenberg CB, Klassen DK, Weir MR, Wiland A, Fink JC, Bartlett ST, Cangro CB, Blahut S, Papadimitriou JC. Islet cell damage associated with tacrolimus and cyclosporine: morphological features in pancreas allograft biopsies and clinical correlation. Transplantation. 1999 Aug 15;68(3):396-402. doi: 10.1097/00007890-199908150-00012. PMID 10459544
- [Result] Terrec F, Jouve T, Naciri-Bennani H, Benhamou PY, Malvezzi P, Janbon B, Giovannini D, Rostaing L, Noble J. Late Conversion From Calcineurin Inhibitors to Belatacept in Kidney-Transplant Recipients Has a Significant Beneficial Impact on Glycemic Parameters. Transplant Direct. 2019 Dec 24;6(1):e517. doi: 10.1097/TXD.0000000000000964. eCollection 2020 Jan. PMID 32047845
- [Result] Rangaswami J, Mathew RO, Parasuraman R, Tantisattamo E, Lubetzky M, Rao S, Yaqub MS, Birdwell KA, Bennett W, Dalal P, Kapoor R, Lerma EV, Lerman M, McCormick N, Bangalore S, McCullough PA, Dadhania DM. Cardiovascular disease in the kidney transplant recipient: epidemiology, diagnosis and management strategies. Nephrol Dial Transplant. 2019 May 1;34(5):760-773. doi: 10.1093/ndt/gfz053. PMID 30984976
- [Result] Anavekar NS, McMurray JJ, Velazquez EJ, Solomon SD, Kober L, Rouleau JL, White HD, Nordlander R, Maggioni A, Dickstein K, Zelenkofske S, Leimberger JD, Califf RM, Pfeffer MA. Relation between renal dysfunction and cardiovascular outcomes after myocardial infarction. N Engl J Med. 2004 Sep 23;351(13):1285-95. doi: 10.1056/NEJMoa041365. PMID 15385655
- [Result] Nankivell BJ, P'Ng CH, O'Connell PJ, Chapman JR. Calcineurin Inhibitor Nephrotoxicity Through the Lens of Longitudinal Histology: Comparison of Cyclosporine and Tacrolimus Eras. Transplantation. 2016 Aug;100(8):1723-31. doi: 10.1097/TP.0000000000001243. PMID 27306529
- [Result] Bertrand D, Terrec F, Etienne I, Chavarot N, Sberro R, Gatault P, Garrouste C, Bouvier N, Grall-Jezequel A, Jaureguy M, Caillard S, Thervet E, Colosio C, Golbin L, Rerolle JP, Thierry A, Sayegh J, Janbon B, Malvezzi P, Jouve T, Rostaing L, Noble J. Opportunistic Infections and Efficacy Following Conversion to Belatacept-Based Therapy after Kidney Transplantation: A French Multicenter Cohort. J Clin Med. 2020 Oct 28;9(11):3479. doi: 10.3390/jcm9113479. PMID 33126667
- [Result] Everly MJ, Roberts M, Townsend R, Bray RA, Gebel HM. Comparison of de novo IgM and IgG anti-HLA DSAs between belatacept- and calcineurin-treated patients: An analysis of the BENEFIT and BENEFIT-EXT trial cohorts. Am J Transplant. 2018 Sep;18(9):2305-2313. doi: 10.1111/ajt.14939. Epub 2018 Jun 16. PMID 29767445
- [Result] Bertrand D, Chavarot N, Gatault P, Garrouste C, Bouvier N, Grall-Jezequel A, Jaureguy M, Caillard S, Lemoine M, Colosio C, Golbin L, Rerolle JP, Thierry A, Sayegh J, Etienne I, Lebourg L, Sberro R, Guerrot D. Opportunistic infections after conversion to belatacept in kidney transplantation. Nephrol Dial Transplant. 2020 Feb 1;35(2):336-345. doi: 10.1093/ndt/gfz255. PMID 32030416
- [Result] Noble J, Jouve T, Janbon B, Rostaing L, Malvezzi P. Belatacept in kidney transplantation and its limitations. Expert Rev Clin Immunol. 2019 Apr;15(4):359-367. doi: 10.1080/1744666X.2019.1574570. Epub 2019 Feb 7. PMID 30676815
- [Result] Noble J, Langello A, Bouchut W, Lupo J, Lombardo D, Rostaing L. Immune Response Post-SARS-CoV-2 mRNA Vaccination in Kidney Transplant Recipients Receiving Belatacept. Transplantation. 2021 Nov 1;105(11):e259-e260. doi: 10.1097/TP.0000000000003923. No abstract available. PMID 34387243
- [Result] Strassl R, Doberer K, Rasoul-Rockenschaub S, Herkner H, Gorzer I, Klager JP, Schmidt R, Haslacher H, Schiemann M, Eskandary FA, Kikic Z, Reindl-Schwaighofer R, Puchhammer-Stockl E, Bohmig GA, Bond G. Torque Teno Virus for Risk Stratification of Acute Biopsy-Proven Alloreactivity in Kidney Transplant Recipients. J Infect Dis. 2019 May 24;219(12):1934-1939. doi: 10.1093/infdis/jiz039. PMID 30668796
- [Result] Doberer K, Haupenthal F, Nackenhorst M, Bauernfeind F, Dermuth F, Eigenschink M, Schiemann M, Klager J, Gorzer I, Eskandary F, Reindl-Schwaighofer R, Kikic Z, Bohmig G, Strassl R, Regele H, Puchhammer-Stockl E, Bond G. Torque Teno Virus Load Is Associated With Subclinical Alloreactivity in Kidney Transplant Recipients: A Prospective Observational Trial. Transplantation. 2021 Sep 1;105(9):2112-2118. doi: 10.1097/TP.0000000000003619. PMID 33587432
- [Result] Sharts-Hopko NC. Hormone replacement therapy and cardiovascular health in midlife women. Medsurg Nurs. 1995 Aug;4(4):314-6. No abstract available. PMID 7627237